CLINICAL TRIAL: NCT00003625
Title: Vincristine, Etoposide and Cyclosporine A in Concert With Standard Dose Radiation Therapy in Diffuse Intrinsic Brain Stem Glioma - A Phase I Study of Dose Escalation of Vincristine
Brief Title: Combination Chemotherapy Plus Radiation Therapy in Treating Patients With Newly Diagnosed Brain Stem Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: 9879; POG-9879; CDR0000066706
Record Dates: First submitted 1999-11-01; First posted 2004-09-13 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Brain Tumors; Central Nervous System Tumors
Keywords: untreated childhood brain stem glioma
MeSH Terms: conditions — Brain Neoplasms; Central Nervous System Neoplasms | interventions — Cyclosporine; Etoposide; Vincristine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stratum 1 (Experimental): Concomitant irradiation and vincristine sulfate in esc dose beginning with 0.8 mg/m2, etoposide and Cyclosporine A given over 6 weeks, then monthly maint courses over 6 mths, with no clinical and radiologic progression. Stable disease indicates continuation of therapy. Clinical deterioration within 4 months of completion of radiation therapy must be confirmed to be PD by imaging. Clinical progression even in the absence of imaging changes will be accepted as reflecting disease progression. Steroids dexamethasone (Decadron) given as clinically indicated and tapered as tolerated. Steroids may decrease capillary permeability to chemotherapeutic agents and antagonise the effect of cyclosporin A. Also contributes to the syndrome of seizures and white matter changes seen with cyclosporine in the post BMT period. If steroid use is required, the recommended schedule of Decadron dosing during the 6 week induction course is 8 mg/m2 divided q 6-8 hours.
  Interventions: Drug: cyclosporine; Drug: etoposide; Drug: vincristine sulfate; Radiation: radiation therapy

INTERVENTIONS:
Drug: cyclosporine
  Other Names: CSA; NSC # 290193
Drug: etoposide
  Other Names: VP-16; VePesid; NSC # 141540
Drug: vincristine sulfate
  Other Names: VCR; Oncovin; NSC # 067574
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining more than one chemotherapy drug with radiation therapy may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combination chemotherapy plus radiation therapy in treating patients with newly diagnosed brain stem glioma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose and dose limiting toxicity of vincristine given as an IV push dose in combination with continuous infusion cyclosporine and oral etoposide concurrent with and prior to radiotherapy in children with newly diagnosed primary intrinsic brain stem glioma. II. Determine the incidence and severity of other toxicities of vincristine in this regimen in these patients. III. Determine a safe and tolerable dose of vincristine under these conditions to be used in phase II studies. IV. Seek preliminary evidence of antitumor activity in this setting in these patients.

OUTLINE: This is dose escalation study of vincristine. Patients receive radiotherapy daily for 6 weeks with concurrent induction chemotherapy. Induction chemotherapy consists of vincristine IV push weekly for 6 weeks, oral etoposide daily on days 1-21 and 29-49 and cyclosporine IV over 2 hours prior to vincristine followed by a continuous 36 hour infusion. Cohorts of 3-6 patients receive escalating doses of vincristine. If dose limiting toxicity (DLT) occurs in 2 or more of 3-6 patients, the maximum tolerated dose (MTD) has been exceeded and the preceding dose is declared the MTD. Maintenance therapy consists of 6 monthly courses of cyclosporine IV over 36 hours beginning on day 1, vincristine IV push on day 1, and oral etoposide daily for days 1-21. Patients are followed every 6 months for 4 years and then annually thereafter.

PROJECTED ACCRUAL: At least 6 patients will be accrued into this study at a rate of 12 patients per year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Newly diagnosed diffuse intrinsic brain stem glioma by MRI Biopsy is neither necessary nor encouraged A least two-thirds of the tumor is in the pons Origin of the tumor is clearly in the pons Must be registered within 28 days of diagnosis Clinical history less than 6 months duration (cranial nerve deficit, long tract signs, or ataxia) No diffuse leptomeningeal disease

PATIENT CHARACTERISTICS: Age: 3 to 21 Performance status: Karnofsky or Lansky 50-100% Life expectancy: At least 6 weeks Hematopoietic: Absolute neutrophil count at least 1,000/mm3 Platelet count at least 75,000/mm3 Hepatic: SGPT less than 2 times normal Renal: Creatinine normal for age OR Creatinine clearance greater than 70 mL/min

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior biologic therapy Chemotherapy: No prior chemotherapy No other concurrent chemotherapy Endocrine therapy: Prior steroids at stable or decreasing doses allowed Radiotherapy: No prior radiotherapy Surgery: Not specified Other: No other concurrent investigational agents

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 1998-12; Primary Completion 2001-02 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Event Free Survival

CONTACTS AND LOCATIONS:
Overall Officials: Mark L. Greenberg, MD, Study Chair — The Hospital for Sick Children
Locations (74):
- United States (65):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of California San Diego Cancer Center, La Jolla, California
  - Lucile Packard Children's Hospital at Stanford, Palo Alto, California
  - Sutter Cancer Center, Sacramento, California
  - Kaiser Permanente-Southern California Permanente Medical Group, San Diego, California
  - Naval Medical Center - San Diego, San Diego, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Nemours Children's Clinic, Jacksonville, Florida
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Walt Disney Memorial Cancer Institute, Orlando, Florida
  - St. Mary's Hospital, West Palm Beach, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - Children's Memorial Hospital, Chicago, Chicago, Illinois
  - Christ Hospital, Oak Lawn, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Via Christi Regional Medical Center-Saint Francis Campus, Wichita, Kansas
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Portland, Maine
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Floating Hospital for Children, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - St. John's Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - University of Missouri-Columbia Hospital and Clinics, Columbia, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University of New Mexico School of Medicine, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Oklahoma Memorial Hospital, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center, Tulsa, Oklahoma
  - Medical University of South Carolina, Charleston, South Carolina
  - James H. Quillen College of Medicine, Johnson City, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Medical City Dallas Hospital, Dallas, Texas
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Baylor College of Medicine, Houston, Texas
  - San Antonio Military Pediatric Cancer and Blood Disorders Center, Lackland Air Force Base, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Clinic, Temple, Texas
  - Vermont Cancer Center, Burlington, Vermont
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Medical School, Charleston Division, Charleston, West Virginia
  - West Virginia University Hospitals, Morgantown, West Virginia
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Canada (6):
  - Alberta Children's Hospital, Calgary, Alberta
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Montreal Children's Hospital, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
  - Centre Hospitalier de L'Universite Laval, Sainte-Foy, Quebec
- Academisch Ziekenhuis Groningen, Groningen, Netherlands
- San Jorge Childrens Hospital, Santurce, Puerto Rico
- Clinique de Pediatrie, Geneva, Switzerland